CLINICAL TRIAL: NCT02217020
Title: A Phase II Study of Neoadjuvant FOLFOXIRI Chemotherapy Alone in Treating Patients With Locally Advanced Rectal Cancer
Brief Title: Neoadjuvant FOLFOXIRI Chemotherapy Alone for Locally Advanced Rectal Cancer
Acronym: FORTUNE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Yanhong Deng, Doctor, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GIHSYSU07
Record Dates: First submitted 2014-08-10; First posted 2014-08-15 (Estimated); Last update posted 2021-04-14 (Actual); Status verified 2021-04

CONDITIONS: Rectal Cancer
Keywords: Rectal Cancer; Locally advanced rectal cancer; Neoadjuvant; chemotherapy; FOLFOXIRI
MeSH Terms: conditions — Rectal Neoplasms | interventions — FOLFOXIRI protocol; Fluorouracil; Oxaliplatin; Irinotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- FOLFOXIRI (Experimental): patients received FOLFOXIRI alone for 4 cycles before surgery.
  Interventions: Drug: FOLFOXIRI

INTERVENTIONS:
Drug: FOLFOXIRI — irinotecan* 165 mg/m² + oxaliplatin 85 mg/m² + leucovorin 200 mg/m² + 5-FU 2800 mg/m² cont. inf. 46h all on day 1 of each 2 weeks cycle
  Other Names: 5-FU; Oxaliplatin; Irinotecan

SUMMARY:
The standard treatment for stage 2/3 rectal cancer is neoadjuvant 5-Fu based chemoradiation. However, preoperative radiation cause kinds of adverse events, some were irreversible. And the survival benefit was not obvious. Whether chemotherapy alone is effective enough in treating rectal cancer is not yet known. Here, the investigators chose all the three active cytotoxic agents (5-FU, Oxaliplatin, Irinotecan) as the neoadjuvant treatment regimen (FOLFOXIRI). The purpose of the study is to evaluate the efficacy of FOLFOXIRI as neoadjuvant regimen in treating patients with locally advanced rectal cancer.

DETAILED DESCRIPTION:
Preoperative chemoradiotherapy could improve the local control of locally advanced rectal cancer, but the role was limited, only 5%. The adverse event cause by radiotherapy was severe. This single phase II trial was aimed to evaluate the efficacy of triplet regimen (FOLFOXIRI) in treating patients with locally advanced rectal cancer. All patients will receive the study regimen every 2 weeks for 4-6 cycles. MRI of the pelvic will be performed after 4 cycles of chemotherapy to assess clinical response. If the tumor response over 20% after 4 cycles of treatment, the patient will go to surgery (TME) directly or 2 more cycles of treatment before surgery under the decision of MDT. On the contrary, if the tumor show poor response (<20%), radiotherapy will be performed before operation. After surgery, 6-8 cycles of mFOLFOX6 will be given as adjuvant chemotherapy.

ELIGIBILITY:
Inclusion Criteria

* Diagnosis of adenocarcinoma of the rectum
* Age: 18-70 years old
* Signed informed consent; able to comply with study and/or follow- up procedures
* Stage of the primary tumor may be determined by ultrasound or MRI
* Stage II (T3-4, N0 [N0 is defined as all imaged lymph nodes < 1.0 cm]) OR stage III (T1-4, N1-2 [with the definition of a clinically positive lymph node being any node ≥ 1.0 cm]
* Tumor palpable by digital rectal exam OR accessible by proctoscope or sigmoidoscope
* Distal border of the tumor must be located < 12 cm from the anal verge
* Tumor amenable to curative resection
* Adequate bone marrow, hepatic and renal function as assessed by the following laboratory requirements conducted within 7 days of starting study treatment:
* Leukocytes ≥ 3.0 x109/ L, absolute neutrophil count (ANC) ≥ 1.5 x109/ L, platelet count ≥ 100 x109/ L, hemoglobin (Hb) ≥ 9g/ dL.
* Total bilirubin ≤1.5 x the upper limit of normal (ULN).
* Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 5 x ULN.
* Alkaline phosphatase limit ≤ 5x ULN.
* Amylase and lipase ≤ 1.5 x the ULN.
* Serum creatinine ≤ 1.5 x the ULN.
* Calculated creatinine clearance or 24 hour creatinine clearance ≥ 50 mL/ min.
* No renal disease that would preclude study treatment or follow-up
* ECOG status: 0～1

Exclusion Criteria:

* Hypersensitivity to fluorouracil, oxaliplatin or irinotecan.
* No More than 4 weeks since prior participation in any investigational drug study
* More than 4 weeks since prior participation in any investigational drug study
* Clear indication of involvement of the pelvic side walls by imaging
* With distant metastasis
* History of invasive rectal malignancy, regardless of disease-free interval
* Fertile patients must use effective contraception
* Uncontrolled hypertension
* Cardiovascular disease that would preclude study treatment or follow-up
* Lack of upper gastrointestinal tract integrity or malabsorption syndrome，active upper gastrointestinal tract bleeding
* Synchronous colon cancer
* Pregnant or nursing, Fertile patients do not use effective contraception
* Other malignancy within the past 5 years except effectively treated squamous cell or basal cell skin cancer, melanoma in situ, carcinoma in situ of the cervix, or carcinoma in situ of the colon or rectum
* No psychiatric or addictive disorders, or other conditions that, in the opinion of the investigator, would preclude study participation
* patients refused to signed informed consent.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2014-08-15; Primary Completion 2016-09-15 (Actual); Study Completion 2017-08-15 (Actual)

PRIMARY OUTCOMES:
The ratio of tumor downstaging to stage 0 and stage I | 2 year
  Tumor downstaging from stage II or III to pathologic complete response (stage 0) and stage I

SECONDARY OUTCOMES:
Average neoadjuvant rectal cancer score | 2 year
  neoadjuvant rectal cancer score (NAR) =[5*pN-3*(cT-pT)+12]^2/9.61 had been proposed and proven to be the surrogate endpoint of overall survival. It refered to the predictive value of lymphnode status and primary tumor downstaging on Overall survival of rectal cancer.
the local Recurrence rate | 3 year
  the ratio of patients with local recurrence within 3 years
Recurrence free survival | 3 years
  3 years recurrence free survival of this group of patients
Reported Adverse events | 2 years
  Number of patients with adverse events and severity according to NCI CTC 4.0 after treatment with this regimen.

CONTACTS AND LOCATIONS:
Locations (1):
- Gastrointestinal Hospital, Sun Yatsen University, Guangzhou, Guangdong, China

REFERENCES:
- [Derived] Zhang J, Li J, Huang M, Xie X, Cai Y, Hu H, Ling J, Wu Z, Deng Y. Neoadjuvant Modified FOLFOXIRI With Selective Radiotherapy in Locally Advanced Rectal Cancer: Long-term Outcomes of Phase II Study and Propensity-Score-Matched Comparison With Chemoradiotherapy. Dis Colon Rectum. 2023 Jul 1;66(7):934-945. doi: 10.1097/DCR.0000000000002424. Epub 2022 Jul 12. PMID 35834598